CLINICAL TRIAL: NCT04347343
Title: Combined Neuromuscular Electrical Stimulation and Blood Flow Restriction Training After Total Knee Arthroplasty
Brief Title: Combined NMES and BFR Training After TKA
Acronym: COMBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Delphi Medical Innovations Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1433
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Total Knee Arthroplasty
Keywords: Blood Flow Restriction; Neuromuscular Electrical Stimulation; BFR; NMES; Rehabilitation
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COMBO (Experimental): Neuromuscular Electrical Stimulation and Blood Flow Restriction (COMBO) in addition to standard postoperative rehabilitation.
  Interventions: Procedure: Standard Rehabilitation + Neuromuscular Electrical Stimulation and Blood Flow Restriction

INTERVENTIONS:
Procedure: Standard Rehabilitation + Neuromuscular Electrical Stimulation and Blood Flow Restriction — Subjects will begin a standardized protocol on post-op day 2. Outpatient visits will be 2x/wk for weeks 0-4 and then 1x/wk for weeks 5-8.
  Subjects will utilize NMES on the quadriceps in the home setting 2x/day for the first 3-4 weeks during isometric contractions at their highest tolerated intensity. Total treatment will begin at 10 minutes.
  At the end of post-op week 2, subjects will be exposed in clinic to BFR on the surgical limb increasing to 80% limb occlusion pressure over weeks 3-4 as tolerated. Initially, BFR and NMES will be performed simultaneously. BFR will then be progressed using active exercises. After completing a safety checklist, subjects will be issued a home BFR unit for use 2x/week (3x total including clinic visit) at which time NMES will be discontinued. BFR exercise intensity will be progressed as tolerated to maintain 20-30% of 1RM.
  Other Names: Blood Flow Restriction; Occlusion Training; BFR; Neuromuscular Electrical Stimulation; NMES

SUMMARY:
The purpose of this feasibility study is to determine the initial efficacy of early combined Neuromuscular Electrical Stimulation (NMES) and Blood Flow Restriction (BFR) in addition to standard rehabilitation in 15 subjects after Total Knee Arthroplasty (TKA). The second aim is to determine the feasibility and patient perceptions of combined NMES and BFR by assessing: 1) adherence, 2) satisfaction and 3) safety.

DETAILED DESCRIPTION:
It's estimated that almost 3.5 million Total Knee Arthroplasties (TKA) will be performed annually by 2030. Despite initiating rehabilitation within 48 hours of surgery, up to a 60% strength loss is noted in the quadriceps one month after TKA. This weakness persists for years after surgery and is associated with decreased gait speed, balance, stair climbing ability and is associated with an increased risk for falls. Approximately 85% of the strength loss after TKA is explained by the combination of voluntary muscle activation deficits and muscle atrophy. Immediately postoperatively, strength loss is primarily due to activation deficits, and as time progresses, muscle atrophy becomes the major contributing factor. Early in the postoperative period, Neuromuscular Electrical Stimulation (NMES) has been shown to diminish activation deficits and improve function after TKA. Blood Flow Restriction (BFR) is a proposed strength training alternative for people who are unable to tolerate traditional strength training at 70-80% of their 1 repetition maximum (1RM), such as those who have just had surgery. Performing low intensity exercise (20-30% of 1RM) with BFR has been shown to achieve similar muscle mass and strength gains when compared to high intensity resistance training. BFR has been studied in people with TKA, but it has been used later in the recovery period (>6 weeks postoperative) when the greatest strength losses have already occurred. The goal of this study is to address both factors of postoperative quadriceps weakness, activation deficit and atrophy, through the use of early NMES and BFR in addition to standard postoperative rehabilitation in an attempt to minimize strength loss and improve functional outcomes.

AIM 1: To determine the initial efficacy of combined neuromuscular electrical stimulation and blood flow restriction training (COMBO) on strength (primary outcome), activation, pain, range of motion, and function compared to historical controls.

Hypothesis 1.1: The COMBO group will have greater attenuation of early postoperative strength losses and improved pain, ROM, and function compared to historical controls.

AIM 2: To determine the feasibility of COMBO by assessing 1) adherence, 2) satisfaction, and 3) safety

Hypothesis 2.1: An 80% adherence rate to the intervention will be observed.

Hypothesis 2.2: Study participants will indicate acceptability of COMBO with a satisfaction survey median score of at least 4/5 ("somewhat satisfied").

Hypothesis 2.3: There will be no intervention-related Adverse Events or Serious Adverse Events during the 8-week protocol.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary unilateral total knee arthroplasty secondary to end-stage osteoarthritis

Exclusion Criteria:

* BMI > 40 kgm2
* Current smoker or history of drug abuse
* Comorbid conditions that substantially limit physical function or would interfere with the participant's ability to successfully complete rehabilitation (e.g. neurologic, vascular, cardiac problems, or ongoing medical treatments)
* Unstable orthopedic conditions that limit function
* Uncontrolled diabetes (hemoglobin A1c level > 8.0)
* Pregnancy
* Preoperative ROM less than 10-120 degrees
* Demand cardiac pacemaker or unstable arrhythmia
* Prior history of DVT/PE
* Thrombophilia or other clotting disorders
* Sickle cell trait/anemia
* History of peripheral vascular disease
* Patient report of easy bruising

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Change in Quadriceps Strength From Baseline to 8 Weeks | Baseline, 4 weeks and 8 weeks after surgery
  Assesses the maximal voluntary isometric contraction strength of the quadriceps muscle using an electromechanical dynamometer.

SECONDARY OUTCOMES:
Change in Quadriceps Activation From Baseline to 8 Weeks | Baseline, 4 weeks and 8 weeks after surgery
  Assesses voluntary activation of the quadriceps using the doublet interpolation technique, where a supramaximal stimulus is applied during a maximal voluntary isometric contraction and again immediately afterward, while the quadriceps muscle is at rest.
Change in Knee Range of Motion (ROM) From Baseline to 8 Weeks | Baseline, 4 weeks and 8 weeks after surgery
  Assesses the mobility of the knee joint. Knee ROM will be measured in the supine position both actively and passively using a long-arm goniometer.
Change in Timed Up and Go (TUG) From Baseline to 8 Weeks | Baseline, 4 weeks and 8 weeks after surgery
  Evaluates mobility through the time required to rise from an arm chair, walk 3 meters, turn and walk back to the arm chair, and return to a seated position.
Change in 30-Second Sit-to-Stand Test (30-STS) From Baseline to 8 Weeks | Baseline, 4 weeks and 8 weeks after surgery
  Assesses lower body strength and the fatigue effect caused by the number of sit-to-stand repetitions that can performed in 30 seconds.
Change in Stair Climbing Test From Baseline to 8 Weeks | Baseline, 4 weeks and 8 weeks after surgery
  Assesses lower body strength, power and balance as measured through the time required to ascend and descend a flight of stairs. Measures a higher level of function that minimizes the possibility of a ceiling effect.
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) From Baseline to 8 Weeks | Baseline, 4 weeks and 8 weeks after surgery
  Assesses self-reported physical function. Scales assess pain, stiffness, and physical function in patients with hip and / or knee osteoarthritis. Total score range is 0-96. Total score is computed by summing three subscales: pain (range 0-20), stiffness (range 0-8), and functional limitations (range 0-68), then dividing by total points possible. Higher scores indicate worse pain, stiffness, and functional limitations.
Adherence to the Intervention as measured by home exercise program logs | 4 weeks and 8 weeks after surgery
  Assesses the adherence of subjects and informs feasibility of intervention. Measured by home exercise program logs.
Satisfaction with Rehabilitation Program as measured by a 5-point Likert scale ranging from "very unsatisfied" to "very satisfied". | 8 weeks after surgery
  Assesses the satisfaction of subjects using a 5-point Likert scale ranging from "very unsatisfied" to "very satisfied" in each of the following rehabilitation program components: overall rehabilitation program, BFR, NMES, and home exercise program. Informs feasibility of intervention.
Safety of COMBO program as measured by adverse events reported per IRB procedures. | 4 weeks and 8 weeks after surgery
  Assess safety of intervention as measured by adverse events related to the COMBO program reported per IRB procedures. Adverse events will be documented at all clinic and testing sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mizner RL, Petterson SC, Stevens JE, Vandenborne K, Snyder-Mackler L. Early quadriceps strength loss after total knee arthroplasty. The contributions of muscle atrophy and failure of voluntary muscle activation. J Bone Joint Surg Am. 2005 May;87(5):1047-53. doi: 10.2106/JBJS.D.01992. PMID 15866968
- [Background] Stevens JE, Mizner RL, Snyder-Mackler L. Quadriceps strength and volitional activation before and after total knee arthroplasty for osteoarthritis. J Orthop Res. 2003 Sep;21(5):775-9. doi: 10.1016/S0736-0266(03)00052-4. PMID 12919862
- [Background] Bade MJ, Kohrt WM, Stevens-Lapsley JE. Outcomes before and after total knee arthroplasty compared to healthy adults. J Orthop Sports Phys Ther. 2010 Sep;40(9):559-67. doi: 10.2519/jospt.2010.3317. PMID 20710093
- [Background] Huang CH, Cheng CK, Lee YT, Lee KS. Muscle strength after successful total knee replacement: a 6- to 13-year followup. Clin Orthop Relat Res. 1996 Jul;(328):147-54. doi: 10.1097/00003086-199607000-00023. PMID 8653948
- [Background] Rantanen T, Guralnik JM, Izmirlian G, Williamson JD, Simonsick EM, Ferrucci L, Fried LP. Association of muscle strength with maximum walking speed in disabled older women. Am J Phys Med Rehabil. 1998 Jul-Aug;77(4):299-305. doi: 10.1097/00002060-199807000-00008. PMID 9715919
- [Background] Skelton DA, Greig CA, Davies JM, Young A. Strength, power and related functional ability of healthy people aged 65-89 years. Age Ageing. 1994 Sep;23(5):371-7. doi: 10.1093/ageing/23.5.371. PMID 7825481
- [Background] Moreland JD, Richardson JA, Goldsmith CH, Clase CM. Muscle weakness and falls in older adults: a systematic review and meta-analysis. J Am Geriatr Soc. 2004 Jul;52(7):1121-9. doi: 10.1111/j.1532-5415.2004.52310.x. PMID 15209650
- [Background] Brown M, Sinacore DR, Host HH. The relationship of strength to function in the older adult. J Gerontol A Biol Sci Med Sci. 1995 Nov;50 Spec No:55-9. doi: 10.1093/gerona/50a.special_issue.55. PMID 7493219
- [Background] Connelly DM, Vandervoort AA. Effects of detraining on knee extensor strength and functional mobility in a group of elderly women. J Orthop Sports Phys Ther. 1997 Dec;26(6):340-6. doi: 10.2519/jospt.1997.26.6.340. PMID 9402571
- [Background] Moxley Scarborough D, Krebs DE, Harris BA. Quadriceps muscle strength and dynamic stability in elderly persons. Gait Posture. 1999 Sep;10(1):10-20. doi: 10.1016/s0966-6362(99)00018-1. PMID 10469937
- [Background] Mizner RL, Petterson SC, Snyder-Mackler L. Quadriceps strength and the time course of functional recovery after total knee arthroplasty. J Orthop Sports Phys Ther. 2005 Jul;35(7):424-36. doi: 10.2519/jospt.2005.35.7.424. PMID 16108583
- [Background] Stevens-Lapsley JE, Balter JE, Wolfe P, Eckhoff DG, Kohrt WM. Early neuromuscular electrical stimulation to improve quadriceps muscle strength after total knee arthroplasty: a randomized controlled trial. Phys Ther. 2012 Feb;92(2):210-26. doi: 10.2522/ptj.20110124. Epub 2011 Nov 17. PMID 22095207
- [Background] Yue C, Zhang X, Zhu Y, Jia Y, Wang H, Liu Y. Systematic Review of Three Electrical Stimulation Techniques for Rehabilitation After Total Knee Arthroplasty. J Arthroplasty. 2018 Jul;33(7):2330-2337. doi: 10.1016/j.arth.2018.01.070. Epub 2018 Feb 6. PMID 29530519
- [Background] Demircioglu DT, Paker N, Erbil E, Bugdayci D, Emre TY. The effect of neuromuscular electrical stimulation on functional status and quality of life after knee arthroplasty: a randomized controlled study. J Phys Ther Sci. 2015 Aug;27(8):2501-6. doi: 10.1589/jpts.27.2501. Epub 2015 Aug 21. PMID 26355656
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Tennent DJ, Hylden CM, Johnson AE, Burns TC, Wilken JM, Owens JG. Blood Flow Restriction Training After Knee Arthroscopy: A Randomized Controlled Pilot Study. Clin J Sport Med. 2017 May;27(3):245-252. doi: 10.1097/JSM.0000000000000377. PMID 27749358
- [Background] Gaunder CL, Hawkinson MP, Tennent DJ, Tubb CC. Occlusion training: pilot study for postoperative lower extremity rehabilitation following primary total knee arthroplasty. US Army Med Dep J. 2017 Jul-Sep;(2-17):39-43. PMID 28853118
- [Background] Kittelson AJ, Stackhouse SK, Stevens-Lapsley JE. Neuromuscular electrical stimulation after total joint arthroplasty: a critical review of recent controlled studies. Eur J Phys Rehabil Med. 2013 Dec;49(6):909-20. Epub 2013 Nov 28. PMID 24285026